CLINICAL TRIAL: NCT04008576
Title: Feasibility of a Group Blended Transdiagnostic Cognitive-behavior Therapy Protocol for the Treatment of Emotional Disorders
Brief Title: Feasibility of a Group Blended Transdiagnostic CBT Protocol for Emotional Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UJaumeI_Transd_Group_Blended
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Anxiety Disorders; Depressive Disorder
Keywords: Transdiagnostic CBT; Internet-delivered CBT; Blended CBT; Group CBT; Negative affect; Positive affect
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Blended Transdiagnostic treatment (Other)
  Interventions: Behavioral: Group Blended Transdiagnostic treatment

INTERVENTIONS:
Behavioral: Group Blended Transdiagnostic treatment — The treatment combines group face-to-face and Internet-delivered psychotherapy: 7 group sessions delivered every 3 weeks plus the use of an online treatment platform between sessions. Its goal is to learn and practice adaptive regulation strategies from a mechanistically transdiagnostic approach, with a focus on both negative and positive affectivity. Each group session will focus on one of the following core components: the first group session will focus on CBT traditional strategies such as motivation for change and psychoeducation about emotions; sessions 2 to 5 will focus on strategies to down-regulate negative affect: present-focused emotional awareness, cognitive flexibility, emotional avoidance and emotion-driven behaviors, and interoceptive and situation-based emotion exposure; session 6 will focus on strategies to regulate positive affect; the final session will teach relapse prevention techniques. All the treatment components are delivered in 16 online treatment modules.

SUMMARY:
The aim of this study is to analyze the feasibility of a blended transdiagnostic group protocol for the treatment of depression and anxiety disorders (emotional disorders) in a one-group clinical trial.

DETAILED DESCRIPTION:
Emotional disorders are the most prevalent mental disorders and they affect the lives of millions of people across the globe. There is an important body of research showing the efficacy of cognitive-behavioral treatments (CBT) for anxiety and depressive disorders (emotional disorders). However, the dissemination and implementation of evidence-based CBT is still one of the principal challenges for research and clinical practice. Over the past two decades, different approaches on how to improve the dissemination and implementation of evidence-based treatments have emerged. In this sense, one important line of research is the transdiagnostic approach to the treatment of emotional disorders. Transdiagnostic treatments "apply the same underlying treatment principles across mental disorders, without tailoring the protocol to specific diagnoses". Broadly, transdiagnostic treatments are based on the premise that the commonalities of psychological disorders outweigh their differences, and that the observed differences (symptoms) are specific manifestations of broader, underlying common psychopathological processes. A number of meta-analyses have shown the efficacy of transdiagnostic treatments. This approach has implications for treatment and clinical practice. For instance, comorbid presentations can be targeted more appropriately, and the costs of training are lower because only one protocol is needed for a range of disorders. Traditionally, transdiagnostic treatments have focused on the regulation of negative affect or neuroticism and less attention has been paid to the regulation of positive affect. However, more recent approaches have emerged that acknowledge the importance of targeting positive affect in addition to negative affect to improve treatment outcomes. Our research group has developed a transdiagnostic protocol that incorporates a component for the regulation of positive affect, with results that support its efficacy in a sample of community patients.

Another approach that could enhance the dissemination and implementation of evidence-based CBT as well as considerably reduce the costs is the use of the Internet to deliver treatments. A number of systematic reviews have shown that Internet-delivered treatments are effective and that they work as effectively as face-to-face psychotherapy. In the context of Internet-delivered treatments, one possibility is the combination of face-to-face and Internet-delivered therapy, also known as blended treatments. The main advantage of blended treatments is its lower cost in comparison with traditional face-to-face psychotherapy. Moreover, blended treatments might be a good alternative for those patients less likely to benefit from guided or unguided Internet-delivered treatments (with no face-to-face contact). On the other hand, group psychotherapy can also help to reduce the costs of therapy. The literature has shown that there are no differences between individual and group CBT for anxiety and depressive disorders.

In spite of the advantages of group CBT, in the specific field of transdiagnostic treatments, research has mainly focused on individual transdiagnostic treatments. Moreover, to our knowledge, no studies have been published that combine blended and group delivery formats to provide transdiagnostic treatments for emotional disorders. The combination of these two treatment approaches to deliver a transdiagnostic treatment might be a highly cost-effective treatment strategy for these disorders. This ultimately could contribute to the dissemination and implementation of evidence-based transdiagnostic CBT.

The goal of this study is to conduct a feasibility trial of a blended transdiagnostic group protocol for the treatment of emotional disorders. The treatment is a transdiagnostic CBT protocol with strategies for the regulation of both negative and positive affectivity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or older
* DSM-5 diagnosis of emotional disorder (panic disorder, agoraphobia, generalized anxiety disorder, social anxiety disorder, major depressive disorder, dysthymic disorder, other specified/unspecified depressive disorder, other specified/unspecified anxiety disorder, obsessive-compulsive disorder)
* Fluent in Spanish
* Daily access to the Internet at home; email address

Exclusion Criteria:

* Diagnosis of a severe mental disorder (schizophrenia, bipolar disorder, substance/alcohol use disorder)
* High risk of suicide
* Receiving another psychological treatment during the study period
* Changes and/or increases in pharmacological treatment during the study period (a decrease is accepted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in the Overall Anxiety Severity and Impairment Scale (OASIS) (Campbell-Sills et al., 2009; González-Robles et al., 2018) at pre-, post-treatment, and at 3-month follow-up. | Pre-treatment, Post treatment (4 months), follow-up (7 months)
  The OASIS is a 5-item self-report scale that evaluates the frequency and severity of anxiety symptoms, the functional impairment related to these symptoms (i.e. school, work, home, or social impairment), and behavioral avoidance. Each item instructs respondents to endorse one of five responses that best describes their experiences over the past week. Response items are coded from 0 to 4, added together to obtain a total score ranging from 0 to 20. Previous studies have shown good internal consistency (α = 0.80), test-retest reliability, and convergent and discriminant validity. The Spanish version has shown good internal consistency (α = 0.86), and convergent and discriminant validity.
Change in the Overall Depression Severity and Impairment Scale (ODSIS) (Bentley et al., 2014; Mira et al., 2019) at pre-, post-treatment, and at 3-month follow-up. | Pre-treatment, Post treatment (4 months), follow-up (7 months).
  The ODSIS is a brief self-reported scale with 5 items that assess the severity and functional impairment associated with depressive symptoms. Items are coded on a 5-point scale (0-4). The sum of the scores is used to obtain the total score, which can be a maximum of 20. The measure has shown excellent internal consistency (α = 0.94 in an outpatient sample, 0.92 in a community sample, and 0.91 in a student sample) and good convergent/discriminant validity. The Spanish validation has excellent internal consistency (α = 0.93), as well as convergent and discriminant validity.

SECONDARY OUTCOMES:
Change in the Positive and Negative Affect Schedule (PANAS) (Watson, Clark, & Tellegen, 1988; Sandín et al., 1999) at pre-, post-treatment, and at 3-month follow-up. | Pre-treatment, Post treatment (4 months), follow-up (7 months).
  The PANAS consists of 20 items that evaluate two independent dimensions: positive affect and negative affect. It contains 10 descriptors evaluating PA (e.g., "enthusiastic," "inspired," "proud") and 10 others assessing NA (e.g., "scared," "irritable," "guilty"). The range for each scale (10 items on each) is from 10 to 50, and the patient has to answer how he or she usually feels regarding each of these emotions. The scale showed excellent internal consistency (α between .84 and .90) and convergent and discriminant validity. The Spanish version has demonstrated good to excellent internal consistency (α = .89 and .91 for PA and NA in women, respectively, and α = .87 and .89 for PA and NA in men, respectively) in college students.
Change in the NEO-five factor Inventory (NEO-FFI) (Costa & McCrae, 1992; Robins, Fraley, Roberts, & Trzesniewski, 2001; Aluja, García, Rossier, & García, 2005) at pre-, post-treatment, and at 3-month follow-up. | Pre-treatment, Post treatment (4 months), follow-up (7 months).
  The NEO FFI is the short version of the NEO-PI-R [88], designed to assess the five personality dimensions through 60 items. In this study, only the subscales of neuroticism and extraversion are used. Each scale contained 12 items with a five-point Likert response format. Two-week retest reliability is uniformly high, ranging from 0.86 to 0.90 for the five scales, and internal consistency ranges from 0.68 to 0.86.The Spanish version of the NEO FFI has been found to be appropriate.
Change in the Quality of Life Index (QLI) (Mezzich, Cohen, Ruiperez, Banzato, & Zapata-Vega, 2011; Mezzich et al., 2000) at pre-, post-treatment, and at 3-month follow-up. | Pre-treatment, Post treatment (4 months), follow-up (7 months).
  The QLI is a self-report questionnaire that consists of 10 items aimed at assessing quality of life in ten areas: psychological well-being, physical well-being, emotional and social support, interpersonal functioning, selfcare and independent functioning, community and service support, occupational functioning, self-realization, spiritual satisfaction, and an overall assessment of quality of life. The Spanish version of the QLI has shown good internal consistency and test-retest reliability in previous studies.
Score on the Work and Social Adjustment Scale (WSAS) (Echezarraga, Calvete, & Las Hayas, 2018; Mundt, Marks, Shear, & Greist, 2002) | Pre-treatment, Post treatment (4 months), follow-up (7 months).
  The WSAS assesses the degree of interference associated with the patients' symptoms in five areas: work, home management, private leisure, social leisure, and family relationships. The questionnaire has 5 items rated on a scale from 0 (not at all) to 8 (very severely). Higher scores indicate greater interference in the different areas.
Score on the Expectations scale and the Opinion scale (adapted from Borkovec & Nau, 1972) | Pre-treatment, post-treatment (4 months).
  Each scale is made up of five items, rated on a scale from 0 (nothing at all) to 10 (completely), that cover how logical the treatment seems to be, to what extent it could satisfy the patient, whether it could be recommended to a person with the same problem, whether it could be used to treat other psychological problems, and its usefulness for the patient's problem. The Expectation scale is applied once the treatment rationale has been explained. Its aim is to measure subjective patient expectations about this treatment. The Opinion scale is administered when the patient has completed the treatment, and its aim is to assess satisfaction with this treatment.
The System Usability Scale (SUS) (Bangor, Kortum, & Miller, 2008; Brooke, 1996) | Post-treatment (4 months).
  The SUS is applied in order to assess the usability of a service or product and the acceptance of technology by the people who use it. The SUS is a simple, ten-item scale that indicates the degree of agreement or disagreement with the statements on a 5-point scale (1=strongly disagree; 5=strongly agree). The final score is obtained by adding the scores on each item and multiplying the result by 2.5. Scores range from 0 to 100, where higher scores indicate better usability.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto González-Robles, Dr, Principal Investigator — Universitat Jaume I; Amanda Díaz-García, Dr, Principal Investigator — Universitat Jaume I
Locations (1):
- University Jaume I, Castellon, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after deidentification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available immediately following publication.
Access Criteria: The data will be available to anyone who wishes to access them.

REFERENCES:
- [Derived] Diaz-Garcia A, Gonzalez-Robles A, Garcia-Palacios A, Fernandez-Felipe I, Tur C, Castilla D, Botella C. Blended transdiagnostic group CBT for emotional disorders: A feasibility trial protocol. Internet Interv. 2021 Jan 7;23:100363. doi: 10.1016/j.invent.2021.100363. eCollection 2021 Mar. PMID 33520670